CLINICAL TRIAL: NCT06830642
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled Study to Assess the Safety, Tolerability and Efficacy of MTR-601, a Novel Oral Treatment in Patients With Cervical Dystonia
Brief Title: Study of the Oral Treatment MTR-601 in Cervical Dystonia
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Pending further safety evaluation
Sponsor: Motric Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MTR-601-201
Record Dates: First submitted 2025-01-31; First posted 2025-02-17 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-12

CONDITIONS: Cervical Dystonia
Keywords: Dystonia; Cervical Dystonia
MeSH Terms: conditions — Torticollis; Dystonia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MTR-601 (Experimental)
  Interventions: Drug: MTR-601
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MTR-601 — Capsule
  Arms: MTR-601
Drug: Placebo — Capsule
  Arms: Placebo

SUMMARY:
Study MTR-601-201 is an 8-week, randomized, placebo-controlled study to examine the safety, tolerability, and efficacy of MTR-601 in participants with cervical dystonia.

DETAILED DESCRIPTION:
Study MTR-601-201 is an 8-week, randomized, placebo-controlled study to examine the safety, tolerability, and efficacy of MTR-601 in participants with cervical dystonia.

Participants will be randomized (1:1) to receive either MTR-601 or matching placebo every day for 4 weeks, after which all participants will be followed for an additional 2 weeks through study treatment washout. The Investigator and Participant will be blinded to the assigned arm. Treatment will be administered via capsules and matching placebo capsules. The total sample size will be approximately 80 participants.

The study will be divided into 3 periods: Screening, Treatment and Follow up.

An initial screening assessment (V1) will occur between Day -90 and Day -2, where individuals will undergo informed consent and have their preliminary eligibility reviewed. Individuals who are found to be eligible will be instructed to not receive their next scheduled botulinum toxin treatment prior to entry into the study.

A full Screening visit (V2) will occur between Day -14 and -1.

Individuals who are confirmed to be eligible after V2, including having not received botulinum toxin treatment for ≥3 months (≥6 months for daxibotulinum ToxinA), will return to clinic on Day 1 for randomization and initiation of study treatment (V3). At this visit individuals will be randomized into the study and receive either MTR-601 or matching placebo to take for the duration of the study and will be discharged home.

Individuals will take the first dose and subsequent doses of study treatment once daily while at home, with weekly visits during the treatment period to assess safety, tolerability and efficacy.

At Day 36 and thereafter, participants may resume treatment with botulinum toxin or daxibotulinum toxinA.

Individuals will return to the clinic 14 days after completion of treatment (Day 42) for the end of study visit (V8) where final safety assessments will be performed. Individuals will then be discontinued from the study.

ELIGIBILITY:
Participants who meet ALL the following inclusion criteria will be eligible to participate in the study:

1. Willing to adhere to study procedures and provide written informed consent prior to the start of any study procedures.
2. Confirmed clinical diagnosis of cervical dystonia with the following:

   * Treatment with botulinum toxin injections (any type) on a stable dosing regimen for ≥ 2 consecutive doses at V2 or a history of botulinum toxin injections within the last 5 years which were discontinued for reasons other than lack of efficacy.
   * 3 months (90 days) since botulinum toxin injection (≥6 months (180 days) for daxibotulinum toxinA) at V3
   * TWSTRS total score ≥ 20 with the following sub scores at V2:
   * Severity ≥ 15
   * Disability ≥ 3
   * Pain score ≥ 1)
   * Willingness to not use botulinum toxin for duration of their study participation
3. Adults 18-80 years of age at the time of consent.
4. Weight ≥40 kg and body mass index (BMI) ≤35 kg/m2.
5. Agree to practice highly effective birth control starting at screening and continuing for 30 days (females) or 90 days (males) after study treatment ends.

   * For females any of the following (no donation of eggs/ova is allowed):
   * Abstinence from heterosexual intercourse.
   * Postmenopausal: absence of menses ≥ 12 months (without an alternative medical condition) and FSH ≥ 40 mIU/mL at screening.
   * Surgically sterile: bilateral oophorectomy, salpingectomy, tubal ligation, or hysterectomy ≥180 days prior to screening.
   * Contraceptive implant or intrauterine device.
   * For males any of the following:
   * Abstinence from heterosexual intercourse.
   * Male condom with spermicide or male condom with vaginal spermicide (gel, foam, or suppository).
   * Surgically sterile: post vasectomy or bilateral orchiectomy ≥180 days prior to screening.
   * No donation of sperm is allowed

Participants who meet ANY of the following criteria will be excluded from participation in the study:

1. History of, or physical examination findings indicating, clinically significant endocrine, neurological, gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, genitourinary, or muscle abnormalities or diseases that, in the opinion of the Investigator, renders the participant unsuitable for the study.
2. History of any of the following:

   * Cervical dystonia due to trauma
   * Chronic contractures in the head and neck musculature
   * Generalized dystonia of any type
   * Myasthenia gravis (MG) or amyotrophic lateral sclerosis (ALS)
3. Use of the following treatment for cervical dystonia:

   * Botulinum toxin (of any type) within 3 months (90 days) (6 months (180 days) for daxibotulinum toxinA) at Baseline (V3)
   * Baclofen by intrathecal pump within 6 months (180 days) months at Baseline (V3)
   * Any previous history of deep brain stimulation or surgery intended to treat or correct cervical dystonia (e.g. myectomy)
   * Other treatments for cervical dystonia (anti-cholinergic, muscle relaxants such as flexeril or oral baclofen, or benzodiazepines) are allowed if the dose has been stable for ≥3 months (90 days).
4. Use of the following medications within 2 weeks prior to V3:

   * CYP3A inhibitors, inducers and substrates.
   * BCRP substrates: rosuvastatin, sulfasalazine
5. Use of the following food or beverages which might interact with MTR-601 within the last week prior to V3:

   - Grapefruit juice or food products containing Seville orange extract (e.g. British orange marmalade, bitter orange liqueurs)
6. History of significant hypersensitivity, intolerance, or allergy to any drug compound, food, or other substance, that, in the opinion of the Investigator, renders the participant unsuitable for the study.
7. Active neoplastic disease or history of any neoplastic disease within 5 years of screening (except for basal or squamous cell carcinoma of the skin or carcinoma in situ that has been definitively treated with standard of care).
8. Active infection (e.g., sepsis, pneumonia, abscess) or a serious infection (e.g., resulting in hospitalization or requiring parenteral antibiotic treatment) within 6 weeks prior to dosing.
9. History of stomach or intestinal surgery or resection that would potentially alter absorption and/or excretion of orally administered drugs (uncomplicated appendectomy and hernia repair are allowed).
10. Any of the following at screening (V2) (if any of these conditions are found on initial ECG, a repeat

    ECG is allowed in consultation with the medical monitor):
    * QT interval corrected for heart rate using Fridericia's formula (QTcF), QRS duration, PR interval outside of normal limits confirmed by repeat measurement, unless deemed non-clinically significant by PI and agreed by Medical Monitor
    * Findings which would make QTc measurements difficult or QTc data uninterpretable
    * History of additional risk factors for Torsades de Pointes (e.g., heart failure, hypokalemia, family history of long QT syndrome)
11. Positive urine alcohol screen or positive urine drug screen (including amphetamines, cocaine, opiates, or barbiturates), at screening (V2).

    * Benzodiazepines will be allowed if prescribed for cervical dystonia, and on a stable dose for ≥3 months (90 days) at screening (V2).
    * Cannabis use and cannabinoid positive drug screen is allowed.
    * Smoking and cotinine positive screen is allowed.
12. Positive hepatitis panel and/or positive human immunodeficiency virus test at screening (V2).
13. Any of the following laboratory values at screening or on Day -1, as confirmed by 1 repeat if necessary:

    * Hemoglobin <11 g/dL for females, and <12 g/dL for males
    * Absolute neutrophil count (ANC) <1.5 × 109

      /L (<1500/μL).
    * Aspartate aminotransferase (AST), alanine aminotransferase (ALT), gammaglutamyl transferase (GGT), alkaline phosphatase (ALP), or total bilirubin >1.5 × upper limit of normal (ULN) at screening or on Day -1, confirmed by 1 repeat if necessary.
14. Participation in a clinical study involving administration of an investigational drug (new chemical entity) or medical device within the last 90 days or 5 half-lives of the investigational medication, whichever is longer, prior to dosing.
15. Receipt of blood products within 2 months prior to Day -1.
16. Donation of blood (>400 mL) or comparable blood loss (>350 mL) from 3 months prior to screening, plasma donation from 2 weeks prior to screening, or platelets donation from 6 weeks prior to screening.
17. Participants who, in the opinion of the Investigator (or designee; including input from participants' general practitioner, as applicable), should not participate in this study.
18. Participants who are investigational site staff members or directly involved in the conduct of the study and their family members or participants who are employed by the Sponsor.
19. Pregnant or nursing (lactating) females

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-28 (Actual); Primary Completion 2026-07-08 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MTR-601 by the incidents of treatment-related adverse events as assessed by CTCAE v5.0 | Baseline to week 6
  To evaluate the safety and tolerability of MTR-601 in participants with cervical dystonia by the incidents of treatments emergent adverse events
To evaluate the efficacy of MTR-601 in participants with cervical dystonia | Baseline to week 4
  To evaluate the efficacy of MTR-601 in participants with cervical dystonia by Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) overall score change.

SECONDARY OUTCOMES:
To evaluate the plasma concentration of MTR-601 in participants with cervical dystonia overall and by age | Day 14 and Day 28
To evaluate the effect of MTR-601 on Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity sub score | Baseline to week 4
To evaluate the effect of MTR-601 on Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) severity sub score | Baseline to week 2
To evaluate the effect of MTR-601 on Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) pain sub score | Baseline to week 4
To evaluate the effect of MTR-601 on Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) pain sub score | Baseline to week 2
To evaluate the effect of MTR-601 on Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) disability sub score | Baseline to week 4
To evaluate the effect of MTR-601 on Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) disability sub score | Baseline to week 2
To evaluate the effect of MTR-601 on Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) overall score | Baseline to week 2

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Arizona Neuroscience Research, LLC, Phoenix, Arizona
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - Keck Medicine of University of Southern California, Los Angeles, California
  - CenExel Rocky Mountain Clinical Research, Englewood, Colorado
  - Neurology One, Orlando, Florida
  - University of South Florida, Tampa, Florida
  - Emory University, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Michigan State University, Department of Neurology, East Lansing, Michigan
  - Quest Research Institute, Farmington Hills, Michigan
  - University of New Mexico, The Nene and Jamie Koch Comprehensive Movement Disorder Clinic, Albuquerque, New Mexico
  - Albany Medical Center Neurosciences Institute, Albany, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Vanderbilt Neurology, The Vanderbilt Clinic, Nashville, Tennessee
  - Kingfisher Cooperative, LLC, Spokane, Washington
  - West Virginia University Medicine, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No